CLINICAL TRIAL: NCT03097445
Title: Long-term Effectiveness of Mailed Nicotine Replacement Therapy: A 5-year Follow-up
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Canadian Cancer Society (CCS) (Other)
Responsible Party: Principal Investigator, John Cunningham, Senior Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 216-2005
Record Dates: First submitted 2017-03-25; First posted 2017-03-31 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Smoking Cessation
Keywords: Smoking; Nicotine; Nicotine Replacement Therapy; Nicotine Patch; Mass Distribution; Tobacco Control; Cancer Prevention; Randomized Controlled Trial
MeSH Terms: conditions — Smoking Cessation; Smoking | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nicotine Replacement Therapy (Experimental): mailed 5 week course of transdermal nicotine patches
  Interventions: Drug: Nicotine patch
- Control (No Intervention): No intervention control group

INTERVENTIONS:
Drug: Nicotine patch — mailed 5-week course of Habitrol® transdermal nicotine patches
  Other Names: Habitrol® transdermal nicotine patches
  Arms: Nicotine Replacement Therapy

SUMMARY:
This study will perform a 5-year follow-up survey of participants in a randomized controlled trial that evaluated the effectiveness of providing 5 weeks of free NRT (in the form of the nicotine patch) by expedited postal mail without behavioural assistance to regular adult smokers recruited across Canada interested in receiving it (clinicaltrials.gov Identifier: NCT01429129).

DETAILED DESCRIPTION:
Our group recently completed a randomized controlled trial evaluating the efficacy of providing 5 weeks of free NRT (in the form of the nicotine patch) by expedited postal mail without behavioural assistance to regular adult smokers recruited across Canada interested in receiving it (clinicaltrials.gov Identifier: NCT01429129). The findings revealed that the provision of free nicotine patches via mail resulted in more than a doubling of 30-day abstinence quit rates at a six-month follow-up compared to the no intervention control group (7.6% versus 3.0%; odds ratio of 2.65). While this trial provided evidence for the effectiveness of nicotine patches as a tobacco cessation aid in real world settings, the findings speak only to the short-term effectiveness of NRT. As evidence for NRT effectiveness has been largely restricted to a final follow-up of 6-12 months after the start of treatment, and relapse to smoking is known to occur beyond this period, it is important to evaluate whether the net benefit of NRT in naturalistic settings can be maintained long-term.

Employing a survey research call centre, trained interviewers will contact participants in the original randomized controlled trial, 5 years post-enrollment. A total of 924 subjects will be eligible to be contacted, however intent-to-treat analyses will evaluate outcomes based on all 1000 participants randomized to condition in the original trial. In this 5-year follow-up survey, interviewers will first assess participants' smoking status, the number of cigarettes smoked per day and their level of nicotine dependence. Participants reporting not currently smoking will be asked whether they have smoked tobacco, even a puff, in the last 30 days (primary outcome measure: abstinence using 30 day point prevalence), past 6 months (secondary outcome measure: prolonged 6-month abstinence), and since the last follow-up survey (secondary outcome measure: > 4 year continuous abstinence). Interviewers will be blind to experimental condition at the time the primary outcome measure will be assessed. The survey component of the proposed study will be conducted over a 2 year period to coincide with the duration of subject recruitment in the original trial. The primary hypothesis is that subjects who received nicotine patches at baseline will display significantly higher quit rates at the 5-year follow-up as compared to subjects who did not receive nicotine patches at baseline.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Current daily smokers who smoke 10 or more cigarettes per day
* Interested in being involved in a smoking study
* Willing to be interviewed at baseline, 8 weeks and 6 months after
* Willing to provide a saliva sample for cotinine analysis at each time point
* Interest in using nicotine patch to quit smoking
* Intent to use nicotine patch within one week of receiving it
* Willing to have nicotine patch sent to their home

Exclusion Criteria:

* Have a medical condition that would would make participation medically hazardous as determined by the list of contraindications for NRT outlined in the CPS and the NRT package insert
* Pregnant, intending on becoming pregnant, or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2017-06-04 (Actual); Primary Completion 2019-08-22 (Actual); Study Completion 2019-08-22 (Actual)

PRIMARY OUTCOMES:
Smoking Cessation | 5-years post intervention
  self-reported 30-day point prevalence abstinence

SECONDARY OUTCOMES:
Prolonged Abstinence | 5 years post intervention
  self-reported prolonged 6-month abstinence
Continuous Abstinence | 5 years post intervention
  self-reported continuous > 4 years abstinence

CONTACTS AND LOCATIONS:
Overall Officials: John Cunningham, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schell C, Godinho A, Kushnir V, Cunningham JA. To send or not to send: weighing the costs and benefits of mailing an advance letter to participants before a telephone survey. BMC Res Notes. 2018 Nov 15;11(1):813. doi: 10.1186/s13104-018-3920-6. PMID 30442187
- [Derived] Kushnir V, Selby P, Zawertailo L, Tyndale RF, Leatherdale ST, Cunningham JA. Long-term effectiveness of mailed nicotine replacement therapy: study protocol of a randomized controlled trial 5-year follow-up. BMC Public Health. 2017 Jul 18;18(1):28. doi: 10.1186/s12889-017-4586-z. PMID 28720080
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching hospital, fully affiliated with the University of Toronto, and a PAHO/WHO Collaborating Centre — http://www.camh.net/research